CLINICAL TRIAL: NCT05791786
Title: The Establishment of a Registry and a Biorepository of Patients With Suspected Amniotic Fluid Embolism (AFE)
Acronym: AFE
Status: Recruiting | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Amniotic Fluid Embolism (AFE) Foundation (Unknown)
Responsible Party: Principal Investigator, Irene Stafford, Associate Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-21-1004
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Amniotic Fluid Embolism
MeSH Terms: conditions — Embolism, Amniotic Fluid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Biospecimen Retention: Samples Without DNA — Maternal blood, umbilical cord blood, and neonatal samples:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AFE: participants of the AFE registry and biorepository include affected individuals diagnosed with AFE
  All subjects or their next of kin must be able to provide a signed and dated informed consent form.
  In the case of lethal AFE, the surviving family member or next of kin must be able to provide a signed and dated informed consent form with an accompanying death certificate and proof of legal kinship
  Interventions: Other: Patient

INTERVENTIONS:
Other: Patient — affected individuals diagnosed with AFE

SUMMARY:
To establish a clinical registry of suspected cases of AFE. The existing registry will be migrated to a new platform,

DETAILED DESCRIPTION:
The registry and the biorepository have prospective and retrospective components.

The prospective component of the registry and the biorepository focuses on the collection of demographic, clinical, and biological material of patients prospectively identified as having the AFE syndrome, including the collection of future samples from survivors and related individuals. Typically, healthcare providers, family members of an affected patient, or patients themselves contact the AFE Foundation. The AFE Foundation provides information about the natural history of the syndrome and its outcomes and invites patients to participate in the registry and biorepository. The AFE Foundation obtains informed consent from patients or next of kin for enrollment in this observational study. There is no randomization or placebo group for this registry as it is exclusively an observational study. If maternal specimens are available pre- and post-event during the hospital admission for delivery, these samples will also be collected from each patient. The only group assignment will be the subjects with a diagnosis of AFE and the subjects' family members including the partner(s) and child (children).

The retrospective component of the registry consists of obtaining clinical information and biological material from patients who have been previously affected by the AFE syndrome. This objective includes obtaining medical records, patient-provided information, pathology reports, autopsy reports, and tissue blocks. Biological samples can also be obtained from survivors and relatives to determine whether there are biomarkers in previously affected patients or whether biomarkers can be elicited from the stimulation of peripheral blood cells. In addition to collecting data and specimens from the patients that are consented and enrolled through the registry, a query of all maternal deaths within 24 hours of birth between 1/2012 to 1/2023 will be performed at the Hermann Hospital system to identify if any of these deaths occurred secondary to AFE. The investigators intend to perform a detailed chart review and collect otherwise discarded tissue if available from the respective hospital to perform special immunohistochemistry staining among women who underwent autopsy.

ELIGIBILITY:
Inclusion Criteria for participants of the AFE registry and biorepository include affected individuals diagnosed with AFE (see below).

* All subjects or their next of kin must be able to provide a signed and dated informed consent form.
* In the case of lethal AFE, the surviving family member or next of kin must be able to provide a signed and dated informed consent form with an accompanying death certificate and proof of legal kinship.
* Participants are expected to be willing to permit collection of data about their affected pregnancy, previous and future pregnancies, and their current and future health conditions.
* Providing biological samples is not required for enrollment.
* Any maternal death in the Hermann Hospital System suspected of having an AFE within 24 hours of childbirth between 1/2012 and 1/2023 will also be included for data analysis and biospecimen studies
* Medical records will be abstracted into a comprehensive case report form and then reviewed by a team of three experts with consensus to determine case classification of three categories, according to criteria previously reported and based on data generated from the previously existing registry:

  (1) Classic AFE is defined by the following indicators:
* Acute hypotension or cardiac arrest,
* Acute hypoxia, defined as dyspnea, cyanosis, or respiratory arrest,
* Coagulopathy, defined as laboratory evidence of intravascular consumption or fibrinolysis or severe clinical hemorrhage in the absence of other explanations,
* Onset of the above during labor, cesarean section, or dilation and evacuation or within 30 minutes post-partum, and
* Absence of any other significant confounding condition or potential explanation for the signs and symptoms observed.

  (2) Not AFE:
* Anything that clinically appears to be a likely result of another pathophysiology, e.g., delayed treatment of postpartum hemorrhage from uterine atony.

  (3) Atypical AFE:
* Subjective determination by the chart reviewer that lies between "classic" and "not," e.g., the patient presents some of the registry criteria and no other explanation.

  (4) Indeterminate: There is not sufficient information to classify in 1-3 above.

The classification of AFE is for research purposes only.

Exclusion Criteria:

* The inability of an individual to provide a signed and dated informed consent form or those who do not wish to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant and postpartum women, survivors, offspring, and relatives of patients with suspected AFE through enrollment or chart review.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2031-10-01 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
To establish a clinical registry of suspected cases of AFE | 1 year
  The existing registry will be migrated to a new platform, thus to enhance and strengthen the content and the quality of the data obtained.
The existing registry will be migrated to a new platform, thus to enhance and strengthen the content and the quality of the data obtained. | 2 weeks
  biological materials would be sought from mothers, their children, and other related individuals
To obtain clinical data and biological specimens from individuals previously enrolled in the registry | 3 weeks
  This objective includes the review of autopsy material and pathology reports, as well as the collection of biological material of survivors and members of the family, to determine whether there is a susceptibility to the AFE syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Irene Stafford, MD, Principal Investigator — UT Health Science Center Health Science Center
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No